CLINICAL TRIAL: NCT03348345
Title: Efficacy of Eat Breathe Thrive, a Yoga-Based Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Give Back Yoga Foundation (Other); Eat Breathe Thrive (Unknown); State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Catherine Cook-Cottone, Principal Investigator, University at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: EBTC01
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2020-09

CONDITIONS: Eating Disorder Symptom
Keywords: eating disorders; prevention; yoga; mindfulness; embodiment; self-regulation; functional action; interoceptive awareness
MeSH Terms: conditions — Feeding and Eating Disorders; Self-Control

STUDY DESIGN:
Intervention Model Description: A computer system will randomly select 100 participants (from 200) to be enrolled in the Eat Breathe Thrive (EBT) intervention group (once a week for two hours) and the other 100 will be wait-listed (WL) for seven weeks. Assessments will be done at week 1 and week 7. At week 7, WL will be enrolled in the 7-week Eat Breathe Thrive program. A second post-test will be given at the end of the second round of Eat Breathe Thrive, administered to those 100 participants only. There will also be three month follow up for all 200 participants.
Masking Description: A computer system will randomly select participants to be enrolled in the program or waitlisted at both time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eat Breathe Thrive Intervention (Experimental): A manualized program designed to prevent eating disorders using psychoeducation, group work, and yoga.
  Interventions: Behavioral: Eat Breathe Thrive
- Wait-List (No Intervention): Participants are placed on a wait-list receiving no intervention.

INTERVENTIONS:
Behavioral: Eat Breathe Thrive — Eat Breathe Thrive (EBT) program which was designed to increase positive body image, awareness, self-regulation, and mindful eating habits. This program aims to achieve these things through psychoeducation of cultural influences of beauty standards, the basic neuropsychological systems in the body and how they affect eating habits, creating a community within the group members for support, and finally through the practice of yoga.
  Arms: Eat Breathe Thrive Intervention

SUMMARY:
The purpose of this study is to evaluate the efficacy of the 7-week Eat Breathe Thrive (EBT) program which was designed to increase positive body image, awareness, self-regulation, and mindful eating habits. This program aims to achieve these things through psychoeducation of cultural influences of beauty standards, the basic neuropsychological systems in the body and how they affect eating habits, creating a community within the group members for support, and finally through the practice of yoga. In this randomized-controlled trial (RCT), investigators will be looking at whether EBT is effective in a community sample of adult (18-65 years old) men and women at preventing and decreasing eating disorder risk and increasing positive body image and emotion regulation skills through being in tune with one's own body, mind, and community. This will take place in a sample of community members taken at ten different sites around the United States and the United Kingdom.

DETAILED DESCRIPTION:
Background: Eating disorders appear predominantly in three types; Anorexia Nervosa [AN]. Bulimia Nervosa [BN], and Binge Eating Disorder [BED]. All three are complex, dangerous mental disorders which deeply affect the quality of life and well-being of the person struggling with it. Eating disorders often sprout from difficulty regulating oneself, and presents as a disturbance of both body image, eating behaviors, and relationship to themselves and others. Since these disorders cause deep disruption between the body and the mind of the person affected, it is imperative that a mind-body approach be taken into consideration for both prevention and treatment options. Likewise, interpersonal relationships are known to suffer as a result of eating disorder symptomatology, and as such, increasing positive social interaction and closeness through community building can act as a support for those affected by this illness. Combining a focus of oneself within support system is one way eating disorders can be healed and even prevented. Since eating disorders are lethal illnesses, prevention of development should be investigated. With a focus on self and body acceptance, community support, and psychoeducation into eating disorders and possible causes, prevention methods can flourish. The Eat Breathe Thrive program has been utilized in communities, eating disorder clinics, and school systems with positive expressed outcomes. Participants in these populations have reported benefits of feeling more empowered, more connected to themselves and others, and more aware of their body's responses to media's attempts at conveying cultural beauty standards. Eat Breathe Thrive aims to accomplish these benefits through community building within a group atmosphere, as well as through yoga, which has been used in the past as an eating disorder prevention and recovery tool via the mind-body connection. By incorporating mind-body practices such as yoga into a program that emphasizes community, self-acceptance, and cultural influence awareness, Eat Breathe Thrive is able to lower eating disorder risk among many populations. From engaging with others and developing a strong investment in themselves, the individuals are then able to sustain proper health, relationships, and overall well-being.

The study will utilize self-report surveys to examine the preventative effects of participation in EBT, a 7-week course, utilizing a randomized-controlled trial (RCT) with a community sample of adult (18-65 years old) men and women.

It is hypothesized that: 1) intervention groups will show a decrease in eating disorder symptoms when compared to controls, 2) intervention groups will show increased in self-care behaviors compared to controls, 3) intervention groups will show an increase in measures of embodied intimacy and a decrease in social and emotional intimacy when compared to controls, 4) intervention groups will show an increase in interoceptive awareness and mindful eating when compared to controls, 5) intervention groups will show a decrease in difficulties with emotion regulation and an increase in distress tolerance when compared to controls, 6) intervention groups will show an increase in their overall mental health functioning, 7) those who are enrolled in two consecutive EBT groups will show better maintenance of increased wellbeing as well as better maintenance in decreased symptomatology as compared to those who took the intervention only one time.

Data will be collected from ten sites around the United States and the United Kingdom where certified Eat Breathe Thrive community facilitators teach the program. Since each group is ran by two facilitators, each group will be recruiting twenty individuals (ten per facilitator) from the community for their respective program for a total of 200 participants. According to calculations of a power analysis, a minimum sample size of 114 participants is required. Given that the average number of participants enrolled in EBT groups is 10-20, investigators believe the sample size of 200 to be attainable across the 10 sites. Each EBT facilitator will recruit at a rate of ten or more participants, resulting in twenty to thirty per group so that each group has at least twenty participants after they are randomized. These participants will be screened by research assistant and doctoral student Esther Estey, to ensure they meet the inclusion criteria and have been deemed eligible to participate in the EBT program by EBT facilitators.

Setting: The facilities in which research will be conducted include the University at Buffalo, yoga studios, and community centers. All locations will be private and confidential.

Data Collection:

* Participants will be assessed at pre-post, and at three month follow up
* Participants will be assessed daily through a phone app for Ecological Momentary Assessments (EMAs)
* Facilitators will complete a Treatment Integrity Check and submit attendance online once per week to maintain adherence to treatment and program protocols and standards. The treatment integrity check will be scored yes or no for a total score for the group.

Data Management and Statistical Analysis: Investigators will use a pretest-posttest randomized control group design. Only quantitative data will be provided for analysis. Specifically, responses on assessment measures, completed at pre- and post-test will be analyzed using a statistical analysis program such as SPSS. All data collected from the online surveys will be screened, checked for outliers, missing data, and other issues. Appropriate techniques will be used for missing data depending on the patterns and frequency (e.g. multiple imputation). Descriptive statistics will be calculated to determine the transfer of Eat Breathe Thrive curriculum concepts from the course into the lives of the participants. An analysis of variance will help in determining whether the Eat Breathe Thrive program had improved outcome results compared to the controlled group at the end of the program and 3 months following program completion.

Quality Assurance: The lead investigator will provide updated copies of all forms (IRB approval, consent forms, protocol, and HIPPA authorization) to each site. There will be weekly contact with each site in order to maintain consistency and support throughout the duration of the study. These check-ins will be done by the lead investigator herself, or two of the Master's level research assistants. All facilitators of groups will complete weekly integrity measures online after every EBT session via email link sent out by research assistant in order to maintain compliance to study protocol. Facilitators will be available for bi-weekly individual phone meetings as well as bi-weekly online group conference calls (through Zoom, which is HIPAA compliant, or other HIPAA compliant web formats). Other forms of bi-weekly communication may include email, text, or other technological means.

Plan to Address Missing Data: Quantitative data (pre and post) will be collected using an online data management software (e.g., SelectSurvey.Net). Access to the researchers' account is secure with a password shared only by lead study researchers. Data will be screened for outliers, suspect patters, or any anomalies in the data set. Dr. Guyker will oversee this and research members will use appropriate techniques to correct and/or work with missing data (e.g. multiple imputation).

Provisions to Monitor Data and Ensure Safety of Subjects: Any evidence that a participant may be at imminent risk (e.g., suicidality, self-harm), whether expressed during the program or upon completing measures, will be immediately addressed by the group facilitators and/or researchers. Specific to facilitators, participants exhibiting these behaviors will be referred, by a their facilitator, to a local treatment provider according to EBT protocol and dismissed from the EBT program as well as discontinued from the study as to protect from further harm. Facilitators will abide by EBT protocol for ensuring safety of participants and withdrawing participants who pose risk to the group. Investigators will survey the data the week after data collection at each assessment point (pretest, posttest 1, posttest 2, and follow-up. If investigators notice any patterns where it might be indicative of the participant needing extra support, investigators will notify the appropriate facilitator to do a referral. The PI and doctoral student Esther Estey will meet and evaluate the data set, watching for trends that are concerning. Although investigators will not be assessing for suicidality and danger to others, investigators will report to facilitators if they notice any general trends that suggest that a participant might need support. The facilitator will then follow up with the participant and provide a referral as indicated.

ELIGIBILITY:
Inclusion Criteria:

* Those included will be men and women between the ages of 18 and 65 who are not pregnant, are willing to sign the consent form, are English-speakers, have not taken EBT before, and have been deemed eligible to participate in the EBT program by EBT facilitators.

Exclusion Criteria:

* Since the scope of this study is adult, non-pregnant English-speaking adults, those excluded will be men and women who are below 18 years old or above 65, pregnant, unable/refuse to sign the consent form, non-English speakers, have taken EBT before, and whom have been deemed ineligible to participate in the EBT program by EBT facilitators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Ecological Momentary Assessments (EMA's) | 7 weeks
  These questions assess eating disorder symptoms, positive coping, and emotion regulation and are sent randomly to participants' mobile phones up to three questions per day.
Integrity Scale | 7 weeks
  Self-report measure of truth and honesty questions. Participants are asked to indicate in the past week whether it's been very difficult, difficult, neutral, easy, or very easy to be honest in the past week with self and with others (1 = very difficult, 2 = difficult, 3= neutral, 4 = easy, 5 = very easy ) and how honest they've been in the past week with themselves and others (1 = not at all honest (about 0%), 2 = a little honest (about 25% of the time), 3= somewhat honest (about 50% of the time), 4 = quite honest (about 75% of the time), 5 = extremely honest (nearly 100% of the time). Higher scores indicate better outcomes (higher levels of ability to be honest and higher frequencies of being honest).
The PTSD Checklist for DSM-5 (PCL-5) | 7 weeks
  Self-report measure of PTSD symptoms
Functional Appreciation Scale (FAS) | 7 weeks
  Self-report measure of levels of functionality appreciation. Participants are asked to indicate the extent to which they agree with statements on appreciation for the functionality of their body (strong agree, disagree, neither agree nor disagree, agree, or strongly agree). Scores on the seven FAS items are averaged, with higher scores reflecting higher levels of functionality appreciation.
Body Appreciation Scale (BAS) | 7 weeks
  Self-report scale of body appreciation. Scale assesses extent of appreciation for one's body. Responses for 10 items are on a 5-point scale (1 = Never, 5 = Always). Scoring procedure entails averaging participants' responses to Items 1-10. Higher scores indicate higher levels of body appreciation.
Eating Disorder Examination Questionnaire (EDE-Q) | 7 weeks
  Participants are to indicate on how many of the past 28 days have they engaged in eating disordered behaviors (0 = no days, 6 = every day) and to what extent have they experienced eating disordered-related cognitions and emotions (0 = not at all, 6 = markedly). It provides frequency data on key behavioral features of eating disorders in terms of number of episodes of the behavior and in some instances number of days on which the behavior has occurred. It provides subscale scores on the severity of aspects of the psychopathology of eating disorders. Subscales are Restraint, Eating Concern, Shape Concern and Weight Concern. The ratings for the relevant items are added together and the sum divided by the total number of items forming the subscales. Higher scores indicate worse outcomes.
Mindful Self-Care Scale-Short (MSCS-S) | 7 weeks
  The MSCS-S is a 33-item scale that measures the self-reported frequency of behaviors that measure self-care behavior. Subscales are positively correlated with body esteem and negative correlated with substance use and eating disordered behavior. There are six additional clinical questions and two general questions for a total of 42 items. The scale helps identify areas of strength and weakness in mindful self-care behavior and assess interventions that serve to improve self-care. The 6 domains are: physical care, supportive relationships, mindful awareness, self-compassion and purpose, mindful relaxation, and supportive structure. There are also 6 clinical items and 3 general items assessing the individual's general/global practices. Participants are asked to indicate the frequency of their self-care behavior over the past week (how much or how often on a scale of 0= never to 6-7 = regularly). The number of items in each domain are averaged. Higher scores indicate better outcome.
Embodied Intimacy Scale (EIS) | 7 weeks
  The EIS is a 10-item scale that assesses levels of embodied intimacy in relationship with self and others (i.e. body expression, body awareness, ability to communicate through the body, ability to maintain boundaries through physical touch). Range is from 0 = never to 5, always. Items 4, 5, and 6 are reversed scored. To score, items are summed and averaged by total number of items. The higher the score, the higher the level of embodied intimacy.
Social Subscale of the Social and Emotional Loneliness Scale for Adults-Short (SELSA-S) | 7 weeks
  The SELSA-S consists of 15 items assessing social and emotional loneliness. It has a 7-point Likert-type response scale ranging from 1 (strongly agree) to 7 (strongly disagree). There are three subscales: Social, Family, and Romantic. Subscale scores are computed by calculating the mean of subscale item responses. Items 2, 3, 5, 6, 8, 9, 11, 12, and 14 are reversed scored. To compute a total score, items indicated are reversed scored then a total mean is computed. High scores indicate high levels of emotional and social loneliness.
Multidimensional Assessment of Interoceptive Awareness (MAIA) | 7 weeks
  The MAIA is a 32-item self-report measure of interoceptive body awareness. It assesses 8 constructs: Noticing, Non-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness, Self-Regulation, Body Listening, and Trusting. The range is from 0 = never, to 5 = always. Summary Score = sum of subscale scores average of each subscale scores ÷ 5. Reverse-score items are 5, 6, and 7 on Not-Distracting, and items 8 and 9 on Not-Worrying. The higher the score, the higher the levels of interoceptive body awareness.
Mindful Eating Questionnaire (MEQ) | 7 weeks
  Self-report measure of mindful eating
Difficulties in Emotion Regulation Scale (DERS) | 7 weeks
  DERS is a 36-item multidimensional assessment of emotion regulation and dysregulation. Total score is the sum of all subscales. The measure yields a total score as well as scores on six sub-scales: Nonacceptance of emotional responses, Difficulty engaging in Goal-directed behavior, Impulse control difficulties, Lack of emotional awareness, Limited access to emotion regulation strategies, and Lack of emotional clarity. Range is from 0 = never to 5 = always. Higher scores suggest greater problems with emotion regulation.
Distress Tolerance Scale (DTS) | 7 weeks
  DTS is a 15-item assessment of beliefs about feelings of distress. Range is from 1 = strongly agree to 5 = disagree. Item 6 is reverse scored. Subscale scores are the mean of the items. The higher-order DTS is formed from the mean of the four subscales. The higher the score, the more positive the outcome.
Substance Abuse subscale of College Counseling Assessment of Psychological Symptoms (CCAPS) | 7 weeks
  Self-report measure of substance abuse. Range is from "never used" to "used 30-60 days in the past 60 days" to assess alcohol and substance use and on the item concerning drinking, three or fewer to seven or more drinks. The higher the score, the more negative the outcome.
Self-Compassion Scale-Short (SCS-S) | 7 weeks
  The SCS-S scale assesses levels of self-compassion. Range is from 1 = almost never to 5 = almost always. Subscale scores are computed by calculating the mean of subscale item responses. To compute a total self-compassion score, reverse score the negative subscale items - self-judgment, isolation, and over-identification (i.e., 1 = 5, 2 = 4, 3 = 3, 4 = 2, 5 = 1) - then compute a total mean. The higher the score, the higher the level of self-compassion.
Demographic information | 7 weeks
  Questions on demographic information
State-Trait Anxiety Inventory for Adults | 7 weeks
  Self-report measure of anxiety symptoms
Beck's Depression Inventory | 7 weeks
  A self-report measure of depression symptoms
Treatment Integrity | 7 weeks
  A weekly assessment of treatment integrity
Pre-Post Class Questions | 7 weeks
  A weekly assessment of stress, relaxation and embodiment
EBT Program Acceptability and Feasibility Questions | 7 weeks
  Post-test assessment of participants' perceptions of acceptability and feasibility of the EBT program

SECONDARY OUTCOMES:
Program Questions for Post-Test and Follow Up | 7 weeks
  Post-test assessment of other mind-body activities engaged in during time of study
Brief COPE Inventory | 7 weeks
  Description of coping mechanisms during stressful events

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Cook-Cottone, PhD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Data sharing is not included in the IRB.

REFERENCES:
- [Background] Cook-Cottone, C. P. (2006). The attuned representational model for the primary prevention of eating disorders: An overview for school psychologists. Psychology in the Schools, 43, 223-230.
- [Background] Cook-Cottone CP. Incorporating positive body image into the treatment of eating disorders: A model for attunement and mindful self-care. Body Image. 2015 Jun;14:158-67. doi: 10.1016/j.bodyim.2015.03.004. Epub 2015 Apr 15. PMID 25886712
- [Background] Cook-Cottone, C. P., Tribole, E., & Tylka, T. (2013). Healthy eating in schools: Evidenced-based interventions to help kids thrive. Washington, DC: American Psychological Association.
- [Background] McIntosh VV, Bulik CM, McKenzie JM, Luty SE, Jordan J. Interpersonal psychotherapy for anorexia nervosa. Int J Eat Disord. 2000 Mar;27(2):125-39. doi: 10.1002/(sici)1098-108x(200003)27:23.0.co;2-4. PMID 10657886